CLINICAL TRIAL: NCT04261699
Title: One-stage Adjustable Strabismus Surgery Under AIVOC
Acronym: AIVOC
Status: Completed | Type: Observational
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL2019-EL01
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Strabismus; Surgery
Keywords: Adjustable strabismus surgery; Target-controlled infusion of Propofol-Reminfentanyl
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to note that one-stage adjustable surgery can be enough to provide satisfactory results for the correction of strabismus in adults thanks to the use of an anesthesia type AIVOC (Target-controlled infusion of Propofol-Remifentanyl)

DETAILED DESCRIPTION:
Adjustable surgery is a surgical treatment technique for strabismus and oculomotor paralysis well known and widely used around the world. The adjustable surgery is done in 2 steps. The first step, performed under general anesthesia, is practically the same as "classic" strabismus surgery however one or more muscles are fixed by temporary sutures. In a second time once the patient is awake and after a new clinical examination the sutures are adjusted and definitively fixed. The adjustment is sometimes made the same day but more often the day after the first intervention because it requires a state of consciousness close to normal.

Anesthesia type Intravenous Intensity Concentration Anesthesia (AIVOC) allows the realization of a surgery under anesthesia general deep (choice of a cerebral or plasma anesthetic target suitable for surgery) but allows a programmed awakening, very fast in full consciousness, condition of an immediate reliable adjustment practically upon stopping the infusion of the anesthetic agent.

The goal is to present an adjustable surgery technique simplified from a logistical point of view since performed in a single step thanks to the contribution of Intravenous Anesthesia with Concentration Objective (AIVOC) and to show that its results are equivalent to a second deferred time.

ELIGIBILITY:
Inclusion Criteria:

* Patient with medical insurance
* Major patient requiring a strabismus surgery
* Patient who received information about study and not having expressed their opposition to participate in the study

Exclusion Criteria:

* Minor patient
* Patient participation in another interventional study
* Patient having expressed their opposition to participate in the study
* Patient for whom it is impossible to give informed information
* Patient under the protection of justice, under curatorship ou under tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient requiring a strabismus surgery not having expressed their oppostion to participate in the study and eligible for anesthesia of type AIVOC.
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Need for a second adjustement time | The day after the intervention
  Use of a second adjustment time the day after surgery

SECONDARY OUTCOMES:
Digital visual scale to assess pain of patient | Before the intervention, before the intervention and one month after the intervention
  Numeric scale numbered from 0 to 10. 0 : no pain, 10 : worst pain possible
Patient comfort assessment questionnaire | 5 minutes after the end of the intervention
  This is a question to determine the comfort of the patient immediatly after the intervention.
  Very comfortable Comfortable Less comfortable Uncomfortable Very uncomfortable
Patient satisfaction questionnaire | 5 minutes after the end of the intervention
  Numeric scale numbered from 0 to 10. 0 : unsatisfied, 10 : very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Erick LAURENT, MD, Principal Investigator — Clinique Saint Jean, Montpellier
Locations (1):
- Clinique Saint Jean, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris RJ, Luff AJ. Adjustable sutures in squint surgery. Br J Ophthalmol. 1992 Sep;76(9):560-2. doi: 10.1136/bjo.76.9.560. No abstract available. PMID 1420063
- [Background] Hassan S, Haridas A, Sundaram V. Adjustable versus non-adjustable sutures for strabismus. Cochrane Database Syst Rev. 2018 Mar 12;3(3):CD004240. doi: 10.1002/14651858.CD004240.pub4. PMID 29527670
- [Background] Farr AK, Guyton DL. Strabismus after retinal detachment surgery. Curr Opin Ophthalmol. 2000 Jun;11(3):207-10. doi: 10.1097/00055735-200006000-00010. PMID 10977229
- [Background] Garrity JA. The surgical management of Graves' ophthalmopathy. Curr Opin Ophthalmol. 1994 Oct;5(5):39-44. PMID 10150815
- [Background] Strominger MB, Richards R. Adjustable sutures in pediatric ophthalmology and strabismus. J Ophthalmic Nurs Technol. 2000 May-Jun;19(3):142-7. No abstract available. PMID 11249243
- [Background] Strominger MB, Richards R. Adjustable sutures in pediatric ophthalmology and strabismus. J Pediatr Ophthalmol Strabismus. 1999 May-Jun;36(3):112-7; quiz 134-5. doi: 10.3928/0191-3913-19990501-07. No abstract available. PMID 10358813
- [Background] Valles-Torres J, Garcia-Martin E, Fernandez-Tirado FJ, Gil-Arribas LM, Pablo LE, Pena-Calvo P. Contact topical anesthesia versus general anaesthesia in strabismus surgery. Arch Soc Esp Oftalmol. 2016 Mar;91(3):108-13. doi: 10.1016/j.oftal.2015.11.012. Epub 2015 Dec 30. English, Spanish. PMID 26743186
- [Background] Tatham A, Amaya L. Immediate post-operative adjustable suture strabismus surgery using a target-controlled infusion of propofol-remifentanil. Ophthalmologica. 2009;223(3):192-5. doi: 10.1159/000200766. Epub 2009 Feb 10. PMID 19204411
- [Background] Karaba VL, Elibol O. One-stage vs. two-stage adjustable sutures for the correction of esotropia. Strabismus. 2004 Mar;12(1):27-34. doi: 10.1076/stra.12.1.27.29009. PMID 15255366
- [Background] Hakim OM, El-Hag YG, Haikal MA. Strabismus surgery under augmented topical anesthesia. J AAPOS. 2005 Jun;9(3):279-84. doi: 10.1016/j.jaapos.2005.01.005. PMID 15956950
- [Background] Bleik JH, Karam VY. Comparison of the immediate with the 24-hour postoperative prism and cover measurements in adjustable muscle surgery: is immediate postoperative adjustment reliable? J AAPOS. 2004 Dec;8(6):528-33. doi: 10.1016/j.jaapos.2004.08.004. PMID 15616499